CLINICAL TRIAL: NCT01573390
Title: Non Invasive and Non-Contact Dual-modal Imaging Of Tissue Oxygenation and Vascular Reactivity Dynamic Imaging Of Tissue Metabolism and Vascular Function.
Brief Title: Non Invasive and Non-Contact Imaging Of Tissue Oxygenation and Vascular Reactivity
Status: Withdrawn | Type: Observational
Why Stopped: most of the study team left the institution prior to study initiation
Sponsor: Chandan K Sen (Other)
Responsible Party: Sponsor-Investigator, Chandan K Sen, Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2010H0017
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Quantitative Validation of Imaging System
Keywords: Non-invasive; tissue-oxygenation; hyperspectral; CWC imaging system

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — there is no biospecimen collection require in this protocol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy participants.

SUMMARY:
1. Quantitative validation of non-contact oxygenation imaging by the CWC imaging system
2. Quantitative validation of non-contact vascular function imaging by the CWC imaging system
3. Evaluation of the clinical usability of the CWC imaging system for further technology development and engineering improvement

DETAILED DESCRIPTION:
The hyperspectral imaging technique estimates cutaneous tissue oxygenation by illuminating tissue and detecting tissue reflectance at different wavelengths. One major advantage of hyperspectral imaging is non-invasive and non-contact detection of tissue functional properties. The dual-mode imaging system integrates hyperspectral and thermal imaging modalities for simultaneous assessment of cutaneous tissue oxygenation and vascular function. This clinical protocol is defined to validate the CWC system on healthy human subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older
* No history of diabetes.
* No history of vascular disease

Exclusion Criteria:

* Under 18 years of age
* Unable to provide informed consent
* Prisoners
* Current smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Interested healthy volunteers
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Non-Contact Oxygenation Imagiing | 1 year
  Quantitative validation of non-contact oxygenation imaging by the CWC imaging system
Non-Contact Vascular Function Imaging | 1 year
  Quantitative validation of non-contact vascular function imaging by the CWC imaging system

SECONDARY OUTCOMES:
Clinical usability for Comprehensive Wound Centers | 1 year
  Evaluation of the clinical usability of the CWC imaging system for further technology development and engineering improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University., Columbus, Ohio, United States

REFERENCES:
- [Result] Xu RX, Huang K, Qin R, Huang J, Xu JS, Ding L, Gnyawali US, Gordillo GM, Gnyawali SC, Sen CK. Dual-mode imaging of cutaneous tissue oxygenation and vascular function. J Vis Exp. 2010 Dec 8;(46):2095. doi: 10.3791/2095. PMID 21178967
- [Result] Singer AJ, Clark RA. Cutaneous wound healing. N Engl J Med. 1999 Sep 2;341(10):738-46. doi: 10.1056/NEJM199909023411006. No abstract available. PMID 10471461
- [Result] Reiber GE. Diabetic foot care. Financial implications and practice guidelines. Diabetes Care. 1992 Mar;15 Suppl 1:29-31. doi: 10.2337/diacare.15.1.s29. PMID 1559416
- [Result] Broughton G 2nd, Janis JE, Attinger CE. Wound healing: an overview. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):1e-S-32e-S. doi: 10.1097/01.prs.0000222562.60260.f9. PMID 16801750
- [Result] Sen CK. Wound healing essentials: let there be oxygen. Wound Repair Regen. 2009 Jan-Feb;17(1):1-18. doi: 10.1111/j.1524-475X.2008.00436.x. PMID 19152646
- [Result] Leach RM, Treacher DF. Oxygen transport-2. Tissue hypoxia. BMJ. 1998 Nov 14;317(7169):1370-3. doi: 10.1136/bmj.317.7169.1370. No abstract available. PMID 9812940
- [Result] Treacher DF, Leach RM. Oxygen transport-1. Basic principles. BMJ. 1998 Nov 7;317(7168):1302-6. doi: 10.1136/bmj.317.7168.1302. No abstract available. PMID 9804723
- [Result] Chang N, Goodson WH 3rd, Gottrup F, Hunt TK. Direct measurement of wound and tissue oxygen tension in postoperative patients. Ann Surg. 1983 Apr;197(4):470-8. doi: 10.1097/00000658-198304000-00017. PMID 6830354
- [Result] Wilson DF. Oxygen dependent quenching of phosphorescence: a perspective. Adv Exp Med Biol. 1992;317:195-201. doi: 10.1007/978-1-4615-3428-0_20. PMID 1288127
- [Result] Griffiths JR, Robinson SP. The OxyLite: a fibre-optic oxygen sensor. Br J Radiol. 1999 Jul;72(859):627-30. doi: 10.1259/bjr.72.859.10624317. No abstract available.
- [Result] Scheffler A, Rieger H. Clinical information content of transcutaneous oxymetry (tcpO2) in peripheral arterial occlusive disease (a review of the methodological and clinical literature with a special reference to critical limb ischaemia). Vasa. 1992;21(2):111-26. PMID 1621428
- [Result] Barker SJ, Tremper KK. Pulse oximetry: applications and limitations. Int Anesthesiol Clin. 1987 Fall;25(3):155-75. doi: 10.1097/00004311-198702530-00010. PMID 3323062
- [Result] Shah SA, Bachrach N, Spear SJ, Letbetter DS, Stone RA, Dhir R, Prichard JW, Brown HG, LaFramboise WA. Cutaneous wound analysis using hyperspectral imaging. Biotechniques. 2003 Feb;34(2):408-13. doi: 10.2144/03342pf01. PMID 12613264
- [Result] Zweier JL, Thompson-Gorman S, Kuppusamy P. Measurement of oxygen concentrations in the intact beating heart using electron paramagnetic resonance spectroscopy: a technique for measuring oxygen concentrations in situ. J Bioenerg Biomembr. 1991 Dec;23(6):855-71. doi: 10.1007/BF00786005. PMID 1663949
- [Result] Ogawa S, Lee TM, Kay AR, Tank DW. Brain magnetic resonance imaging with contrast dependent on blood oxygenation. Proc Natl Acad Sci U S A. 1990 Dec;87(24):9868-72. doi: 10.1073/pnas.87.24.9868. PMID 2124706
- [Result] Valk PE, Mathis CA, Prados MD, Gilbert JC, Budinger TF. Hypoxia in human gliomas: demonstration by PET with fluorine-18-fluoromisonidazole. J Nucl Med. 1992 Dec;33(12):2133-7. PMID 1334136
- [Result] Hosokawa R, Nohara R, Fujibayashi Y, Okuda K, Ogino M, Hirai T, Fujita M, Tamaki N, Konishi J, Sasayama S. Myocardial metabolism of 123I-BMIPP in a canine model with ischemia: implications of perfusion-metabolism mismatch on SPECT images in patients with ischemic heart disease. J Nucl Med. 1999 Mar;40(3):471-8. PMID 10086713
- [Result] Djordjevich L, Sadove MS. Basic principles of electrohaemodynamics. J Biomed Eng. 1981 Jan;3(1):25-33. doi: 10.1016/0141-5425(81)90101-1. PMID 7464087
- [Result] Kongstad L, Grande PO. The role of arterial and venous pressure for volume regulation of an organ enclosed in a rigid compartment with application to the injured brain. Acta Anaesthesiol Scand. 1999 May;43(5):501-8. doi: 10.1034/j.1399-6576.1999.430503.x. PMID 10341996
- [Result] Whiston R. Wound care. Principles of Doppler. Nurs Times. 1996 May 15-21;92(20):66-70. No abstract available. PMID 8715837
- [Result] Luypaert R, Boujraf S, Sourbron S, Osteaux M. Diffusion and perfusion MRI: basic physics. Eur J Radiol. 2001 Apr;38(1):19-27. doi: 10.1016/s0720-048x(01)00286-8. PMID 11287161
- [Result] Khan F, Newton DJ. Laser Doppler imaging in the investigation of lower limb wounds. Int J Low Extrem Wounds. 2003 Jun;2(2):74-86. doi: 10.1177/1534734603256271. PMID 15866831
- [Result] Hlavova A, Linhart J, Provsky I, Ganz V, Fronek A. Measurement of blood flow in the femoral artery in man at rest and during exercise by local thermodilution. Scand J Clin Lab Invest Suppl. 1967;99:86-9. No abstract available. PMID 4861921
- [Result] Johnson LL, Seldin DW. Clinical experience with technetium-99m teboroxime, a neutral, lipophilic myocardial perfusion imaging agent. Am J Cardiol. 1990 Oct 16;66(13):63E-67E. doi: 10.1016/0002-9149(90)90614-7. PMID 2220625
- [Result] Kupriyanov VV, Nighswander-Rempel S, Xiang B. Mapping regional oxygenation and flow in pig hearts in vivo using near-infrared spectroscopic imaging. J Mol Cell Cardiol. 2004 Nov;37(5):947-57. doi: 10.1016/j.yjmcc.2004.07.007. PMID 15522272
- [Result] Greenman RL, Panasyuk S, Wang X, Lyons TE, Dinh T, Longoria L, Giurini JM, Freeman J, Khaodhiar L, Veves A. Early changes in the skin microcirculation and muscle metabolism of the diabetic foot. Lancet. 2005 Nov 12;366(9498):1711-7. doi: 10.1016/S0140-6736(05)67696-9. PMID 16291064
- [Result] Myers DE, Anderson LD, Seifert RP, Ortner JP, Cooper CE, Beilman GJ, Mowlem JD. Noninvasive method for measuring local hemoglobin oxygen saturation in tissue using wide gap second derivative near-infrared spectroscopy. J Biomed Opt. 2005 May-Jun;10(3):034017. doi: 10.1117/1.1925250. PMID 16229661
- [Result] Khaodhiar L, Dinh T, Schomacker KT, Panasyuk SV, Freeman JE, Lew R, Vo T, Panasyuk AA, Lima C, Giurini JM, Lyons TE, Veves A. The use of medical hyperspectral technology to evaluate microcirculatory changes in diabetic foot ulcers and to predict clinical outcomes. Diabetes Care. 2007 Apr;30(4):903-10. doi: 10.2337/dc06-2209. Epub 2007 Feb 15. PMID 17303790
- [Result] Khoobehi B, Beach JM, Kawano H. Hyperspectral imaging for measurement of oxygen saturation in the optic nerve head. Invest Ophthalmol Vis Sci. 2004 May;45(5):1464-72. doi: 10.1167/iovs.03-1069. PMID 15111603
- [Result] Jarm T, Kragelj R, Liebert A, Lukasiewitz P, Erjavec T, Preseren-Strukelj M, Maniewski R, Poredos P, Miklavcic D. Postocclusive reactive hyperemia in healthy volunteers and patients with peripheral vascular disease measured by three noninvasive methods. Adv Exp Med Biol. 2003;530:661-9. doi: 10.1007/978-1-4615-0075-9_66. PMID 14562764
- [Result] Hueber DM, Franceschini MA, Ma HY, Zhang Q, Ballesteros JR, Fantini S, Wallace D, Ntziachristos V, Chance B. Non-invasive and quantitative near-infrared haemoglobin spectrometry in the piglet brain during hypoxic stress, using a frequency-domain multidistance instrument. Phys Med Biol. 2001 Jan;46(1):41-62. doi: 10.1088/0031-9155/46/1/304. PMID 11197678
- [Result] Franceschini MA, Moesta KT, Fantini S, Gaida G, Gratton E, Jess H, Mantulin WW, Seeber M, Schlag PM, Kaschke M. Frequency-domain techniques enhance optical mammography: initial clinical results. Proc Natl Acad Sci U S A. 1997 Jun 10;94(12):6468-73. doi: 10.1073/pnas.94.12.6468. PMID 9177241